CLINICAL TRIAL: NCT04314570
Title: Saphenous Nerve Block for Post-Op Pain Control After Tibial Plateau ORIF
Brief Title: Saphenous Nerve Block After Tibial Plateau ORIF
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Jean-Louis Horn, Principal Investigator, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 31480
Record Dates: First submitted 2020-03-16; First posted 2020-03-19 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Tibial Plateau Fracture; Pain, Postoperative
MeSH Terms: conditions — Tibial Plateau Fractures; Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ropivacaine Treatment (Experimental): After the patient has been consented for a post-operative nerve block, physicians will provide a loading dose of Ropivacaine through the catheter. After one hour, the patient will receive their Ropivacaine infusions as per standard protocol.
  Interventions: Procedure: Saphenous Nerve Block with Ropivacaine Treatment
- Saline Control (Placebo Comparator): After the patient has been consented for a post-operative nerve block, physicians will provide a loading dose of Normal Saline through the catheter. After one hour, the patient will receive their Ropivacaine infusions as per standard protocol.
  Interventions: Procedure: Saphenous Nerve Block with Saline Control

INTERVENTIONS:
Procedure: Saphenous Nerve Block with Ropivacaine Treatment — Regional Anesthesia nerve blocks have become standard practice for several orthopedic surgeries for post-operative pain management, however concerns for compartment syndrome have prevented nerve blocks to become common practice for tibial plateau open reduction internal fixation pain management. Interestingly, saphenous nerve blocks do not cover the sciatic nerve, allowing for pain management while reducing concerns that it may possibly mask compartment syndrome. Patients will receive ropivacaine through the catheter from the start of the nerve block.
  Arms: Ropivacaine Treatment
Procedure: Saphenous Nerve Block with Saline Control — Regional Anesthesia nerve blocks have become standard practice for several orthopedic surgeries for post-operative pain management, however concerns for compartment syndrome have prevented nerve blocks to become common practice for tibial plateau open reduction internal fixation pain management. Interestingly, saphenous nerve blocks do not cover the sciatic nerve, allowing for pain management while reducing concerns that it may possibly mask compartment syndrome. Patients will receive a loading dose of Normal Saline through the catheter. After one hour, the patient will receive their Ropivacaine infusions as per standard protocol.
  Arms: Saline Control

SUMMARY:
Fractures of the tibial plateau, while very painful, typically do not receive nerve blocks. This is because of a concern that the numbness from a nerve block would "mask" the typically painful symptoms of compartment syndrome, a condition that can lead to a permanent loss of function of the injured limb. Our study aims to evaluate the effectiveness of saphenous nerve block for pain management after surgical repair of a tibial plateau fracture. Based on cadaver studies and our clinical experience, we suspect that the saphenous nerve contributes to pain sensations of the tibial plateau and will not mask the pain from a compartment syndrome. In summary, while saphenous nerve block represents a safe option after tibial plateau open reduction internal fixation (ORIF), we aim to evaluate its effectiveness in this patient population.

ELIGIBILITY:
Inclusion Criteria:

* Tibial plateau fracture presenting for ORIF
* Age greater than or equal to 18 years

Exclusion Criteria:

* Other concomitant life-threatening injuries
* History of chronic pain prior to tibial plateau ORIF
* Age <18 years old
* Pregnancy
* Any condition impairing patient's ability to consent to participation in study
* Existing condition contraindicating a nerve block
* Non-English Speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Pain Scores | Through hospital stay, an average of 3 days
  Pain scores on a scale from 0 to 10 will be collected by the research staff for 1 hour following the post-operative block. Pain scores will also be collected by the nurses throughout the patient's stay.
Opioid requirements | Through hospital stay, an average of 3 days
  Opioid medications recorded in opioid morphine equivalents will be recorded by the research staff for the first hour following the post-operative nerve block. Opioid medications will be collected by the nurses throughout the patient's stay.
Length of Stay | Through hospital stay, an average of 3 days
  The patient's length of stay in the hospital will be collected by the research staff following the patient's discharge.